CLINICAL TRIAL: NCT00155831
Title: Neural Development and Its Influencing Factors in Premature Infants With Chronic Lung Disease
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Suh-Fang Jeng/Director, Professor, School of Psysical Therapy, National Taiwan University
Other Study IDs: 9100208567
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2010-03-31 (Estimated); Status verified 2010-03

CONDITIONS: Premature Birth
Keywords: Premature infants; Kicking; Stepping; Walking; Motor development; Kinematics
MeSH Terms: conditions — Premature Birth; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Current approaches to treatment of premature infants at risk for neurodevelopmental disabilities have emphasized early assessment and intervention within the first year of life to optimize their developmental outcome. However, the information concerning the course of early neuromotor development and the factors contributing to neurodevelopmental disabilities in premature infants with CLD is limited. Therefore, the major purposes of this three-year multi-centered developmental follow-up study are threefold. (1) We will prospectively evaluate the early neuromotor performance of premature infants with CLD and premature infants without CLD from birth until 12 months of corrected age. (2) We will follow up the neurodevelopmental outcome of these infants at 12,18 and 24 months of corrected age to identify the early neuromotor impairments that predict later neurodevelopmental disabilities. (3) We will examine two potential influencing factors i.e., respiratory disease itself and brain lesions that may contribute to the neurodevelopmental disabilities in premature infants with CLD.

DETAILED DESCRIPTION:
In the past three decades, the advancement of perinatal and neonatal care has resulted in a marked improvement in the survival of premature infants. However, this has been offset by an increasing incidence of chronic lung disease (CLD). Longitudinal follow-up studies indicated that premature infants resolving from CLD have a higher risk of neurodevelopmental disabilities and have poorer cognitive performance at school age compared with those without. Current approaches to treatment of premature infants at risk for neurodevelopmental disabilities have emphasized early assessment and intervention within the first year of life to optimize their developmental outcome. However, the information concerning the course of early neuromotor development and the factors contributing to neurodevelopmental disabilities in premature infants with CLD is limited. Therefore, the major purposes of this three-year multi-centered developmental follow-up study are threefold. First, we will prospectively evaluate the early neuromotor performance of premature infants with CLD and premature infants without CLD from birth until 12 months of corrected age. Neuromotor performance will be assessed using the Neonatal Neurobehavioral Examination- Chinese version during neonatal period, and the Alberta Infant Motor Scale and a three-dimensional video motion analysis system during infancy. Secondly, we will follow up the neurodevelopmental outcome of these infants at 12,18 and 24 months of corrected age to identify the early neuromotor impairments that predict later neurodevelopmental disabilities. Neurodevelopmental outcome will be assessed using the Bayley Scale of Infant Development- 2nd edition and physician's neurological diagnosis. Thirdly, we will examine two potential influencing factors i.e., respiratory disease itself and brain lesions that may contribute to the neurodevelopmental disabilities in premature infants with CLD. Respiratory disease will be assessed using the Clinical and Roentgenographic Scoring Systems for Assessing Bronchopulmonary Dysplasia during neonatal period and pulse oximeter during infancy. Brain lesions will be assessed with cranial ultrasonography and magnetic resonance imaging. This research project will enroll 60 premature infants with CLD and 60 premature infants without CLD from National Taiwan University Hospital and MacKay Memorial Hospital. The groups will be matched for birth weight. The results of this study will help understand the course and nature of early neuromotor development in premature infants with CLD. The obtained early neuromotor predictors will assist clinician early detection of infants who are at greatest risk for developmental disabilities and are in most need of early intervention services. The identified factors for adverse neurodevelopment in premature infants with CLD will assist health care professionals in designing prevention and intervention programs to enhance their developmental outcome. Furthermore, the obtained database will help develop a national monitoring system for measuring developmental effects of respiratory management and early intervention programs for premature infants with neonatal respiratory disease.

ELIGIBILITY:
Inclusion Criteria:

* BW below 2,000 gm
* GA under 34 weeks
* Admission to the NICU within the first 7 days

Exclusion Criteria:

* Existence of congenital anomalies and genetic disease

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: premature infants with chronic lung disease(CLD) and 60 premature infants without CLD from National Taiwan University Hospital and MacKay Memorial Hospital
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2003-08; Primary Completion 2005-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suh-Fang Jeng, Sc.D, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Li SJ, Tsao PN, Tu YK, Hsieh WS, Yao NJ, Wu YT, Jeng SF. Cognitive and motor development in preterm children from 6 to 36 months of age: Trajectories, risk factors and predictability. Early Hum Dev. 2022 Sep;172:105634. doi: 10.1016/j.earlhumdev.2022.105634. Epub 2022 Jul 28. PMID 35921693